CLINICAL TRIAL: NCT02527343
Title: A Randomized, Double-Blind, Placebo-Controlled, With an Open Label Extension, Phase 2/3 Study of ISIS 304801 Administered Subcutaneously to Patients With Familial Partial Lipodystrophy
Brief Title: The BROADEN Study: A Study of Volanesorsen (Formerly IONIS-APOCIIIRx) in Participants With Familial Partial Lipodystrophy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study terminated early at a time point when sufficient data had been accumulated to inform a decision on further development of volanesoresen in participants with FPL.
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 304801-CS17; 2015-000493-35 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Familial Partial Lipodystrophy
MeSH Terms: conditions — Lipodystrophy, Familial Partial | interventions — ISIS 304801

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Placebo/Volanesorsen (Experimental): Randomized Period: Volanesorsen-matching placebo as SC, QW for Weeks 1-52. Participants who received volanesorsen-matching placebo in RT period and not enter in OLE period went straight to 13-week PT follow-up period. Dose adjustment based on monitoring rules were allowed.
  OLE Period: Participants who received volanesorsen-matching placebo in RT period and completed RT period, were to receive 300 mg of volanesorsen as SC QW for 52 weeks (Weeks 53-104) in OLE period. Dose adjustment based on monitoring rules were allowed. After Week 104, participants had option of continuing treatment with 300 mg of volanesorsen as SC injection for up to additional 52 weeks (Weeks 105-156). Participants not entered in option for additional 52 weeks of dosing in OLE PT period went straight to 13-week PT follow-up period after completion of first 52 weeks (Weeks 53-104) of OLE. Participants entered in OLE PT period went straight to 13-week PT follow-up period after completion of Week 156 of OLE.
  Interventions: Drug: volanesorsen; Drug: Placebo
- Volanesorsen (Experimental): Randomized Period: 300 mg of volanesorsen as SC, QW for Weeks 1-52. Participants who received 300 mg of volanesorsen in RT period and did not enter in OLE period went straight to 13-week PT follow-up period. Dose adjustment based on monitoring rules were allowed.
  OLE Period: Participants who received volanesorsen in RT period and completed RT period, were to receive 300 mg of volanesorsen as SC QW for 52 weeks (Weeks 53-104) in OLE period. Dose adjustment based on monitoring rules were allowed. After Week 104, participants had option of continuing treatment with 300 mg of volanesorsen as SC injection for up to additional 52 weeks (Week 105-156). Participants who were not entered in option for additional 52 weeks of dosing in OLE PT period went straight to 13-week PT follow-up period after completion of first 52 weeks (Weeks 53-104) of OLE. Participants entered in OLE PT period went straight to 13-week PT follow-up period after completion of Week 156 of OLE.
  Interventions: Drug: volanesorsen

INTERVENTIONS:
Drug: volanesorsen — 300 mg of volanesorsen administered subcutaneous (SC) injection, once-weekly (QW).
  Other Names: ISIS 304801; IONIS-APOCIIIRx
Drug: Placebo — Volanesorsen-matching placebo administered SC injection.
  Arms: Placebo/Volanesorsen

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of volanesorsen given for 52 weeks in a randomized treatment (RT) period in participants with familial partial lipodystrophy (FPL). Following the randomized treatment period, participants who did not enter the open-label extension (OLE) period went straight to the 13-week post-treatment (PT) follow-up period and participants who were entered in the OLE period continued to receive volanesorsen for another 52 weeks (Weeks 53 to 104). Following the Week 104 visit of the OLE period, participants had an option of continued dosing for up to an additional 52 weeks (Week 105 to 156). Participants who did not enter the OLE period went straight to a 13-week post-treatment follow-up period. Following the Week 104 OLE period, participants were entered a 13-week post-treatment follow-up period, if they did not choose the option for continued dosing.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law.
* Clinical diagnosis of familial partial lipodystrophy (FPL) plus diagnosis of type 2 diabetes mellitus, hypertriglyceridemia, and fatty liver.
* Diagnosis of FPL is based on deficiency of subcutaneous body fat in a partial fashion assessed by physical examination and low skinfold thickness in anterior thigh by caliper measurement: men (less than or equal to [≤] 10 millimeters [mm]) and women (≤ 22 mm), and at least 1 of the following:

  1. Genetic diagnosis of FPL OR
  2. Family history of FPL or of similar abnormal fat distribution plus 1 Minor Criteria OR
  3. In the absence of FPL-associated genetic variant or family history, 2 Minor Criteria and body mass index (BMI) less than (<) 35 kilogram per meter square (kg/m^2).
* Diabetes not well controlled on antidiabetic therapy with glycated hemoglobin (Hb) HbA1c more than or equal to (≥) 7 percentage (%) to ≤ 12% at Screening.
* Hypertriglyceridemia with fasting triglycerides (TG) levels greater than or equal to (≥) 500 milligrams per deciliter (mg/dL) (≥ 5.7 millimoles per liter [mmol/L]) at Screening and Qualification visit, or Fasting TG levels ≥ 200 (≥ 2.26 mmol/L) at both Screening and Qualification Visits for participants who meet the genetic or family history criteria.
* Presence of hepatosteatosis (fatty liver), as evidenced by a screening magnetic resonance imaging (MRI) indicating a hepatic fat fraction (HFF) ≥ 6.4%.

Exclusion Criteria:

* A diagnosis of generalized lipodystrophy.
* A diagnosis of acquired partial lipodystrophy.
* Acute pancreatitis within 4 weeks of Screening.
* History within 6 months of Screening of acute or unstable cardiac condition.
* Low-density lipoprotein cholesterol (LDL-C) more than (>) 130 mg/dL on maximal tolerated statin therapy.
* Platelet count < lower limit of normal (LLN).
* Treatment with metreleptin within the last 3 months prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - IONIS Investigative Site, Ann Arbor, Michigan
  - IONIS Investigative Site, Rochester, Minnesota
  - IONIS Investigative Site, St Louis, Missouri
  - IONIS Investigative Site, Morehead City, North Carolina
  - IONIS Investigative Site, Philadelphia, Pennsylvania
  - IONIS Investigative Site, Dallas, Texas
- IONIS Investigative Site, Leuven, Belgium
- IONIS Investigative Site, Rio de Janeiro, Brazil
- IONIS Investigative Site, Halifax, Nova Scotia, Canada
- IONIS Investigative Site, Münster, Germany
- IONIS Investigative Site, Amsterdam-Zuidoost, Netherlands
- IONIS Investigative Site, Moscow, Russia

REFERENCES:
- [Derived] Prohaska TA, Alexander VJ, Karwatowska-Prokopczuk E, Tami J, Xia S, Witztum JL, Tsimikas S. APOC3 inhibition with volanesorsen reduces hepatic steatosis in patients with severe hypertriglyceridemia. J Clin Lipidol. 2023 May-Jun;17(3):406-411. doi: 10.1016/j.jacl.2023.04.007. Epub 2023 Apr 27. PMID 37164837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 study centers in the United States, Russia, Brazil, Germany, Belgium, Canada, and Netherlands from 28 December 2015 to 13 November 2019.
Pre-assignment Details: A total of 40 participants were randomized into this study.
Groups:
- Randomized Treatment Period: Placebo: Participants received volanesorsen-matching placebo as a subcutaneous (SC) injection once-weekly from Weeks 1 to 52 of the randomized treatment (RT) period. Participants were allowed dose adjustment based on monitoring rules.
- Randomized Treatment Period: Volanesorsen: Participants received 300 mg of volanesorsen as a SC injection once-weekly from Weeks 1 to 52 of the randomized treatment period. Participants were allowed dose adjustment based on monitoring rules.
- Randomized Post-Treatment Follow-up Period: Placebo: Following the randomized treatment period, participants who received volanesorsen-matching placebo in randomized treatment period and did not enter the open-label extension (OLE) period went straight to the 13-week post-treatment (PT) follow-up period.
- Randomized Post-Treatment Follow-up Period: Volanesorsen: Following the randomized treatment period, participants who received 300 mg of volanesorsen in randomized treatment period and did not enter in the OLE period went straight to the 13-week post-treatment follow-up period.
- Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen: Participants in the Randomized Treatment Period: Placebo arm group who completed the randomized treatment period, were to receive 300 mg of volanesorsen as a SC injection once-weekly for 52 weeks (from Weeks 53 to 104) in the OLE period. Participants were allowed dose adjustment based on monitoring rules. After Week 104 of the OLE period, participants had the option of continuing treatment with 300 mg of volanesorsen as a SC injection for up to an additional 52 weeks (from Week 105 to 156). Participants who were not entered in the option for an additional 52 weeks of dosing in the OLE post-treatment period went straight to a 13-week post-treatment follow-up period after completion of the first 52 weeks (from Weeks 53 to 104) of the OLE. Participants who were entered in the OLE post-treatment period went straight to a 13-week post-treatment follow-up period after completion of Week 156 of the OLE.
- Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen: Participants in the Randomized Treatment Period: Volanesorsen arm group who completed the randomized treatment period, received 300 mg of volanesorsen as a SC injection once-weekly for 52 weeks (from Weeks 53 to 104) in the OLE period. Participants were allowed dose adjustment based on monitoring rules. After Week 104 of the OLE period, participants had the option of continuing treatment with 300 mg of volanesorsen as a SC injection for up to an additional 52 weeks (from Week 105 to 156). Participants who were not entered in the option for an additional 52 weeks of dosing in the OLE post-treatment period went straight to a 13-week post-treatment follow-up period after completion of the first 52 weeks (from Weeks 53 to 104) of the OLE. Participants who were entered in the OLE post-treatment period went straight to a 13-week post-treatment follow-up period after completion of Week 156 of the OLE.
Period: RT Period: Weeks 1 to 52
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen | Randomized Post-Treatment Follow-up Period: Placebo | Randomized Post-Treatment Follow-up Period: Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen
Started | 19 | 21 | 0 | 0 | 0 | 0
Completed | 13 | 14 | 0 | 0 | 0 | 0
Not Completed | 6 | 7 | 0 | 0 | 0 | 0
Not completed — Investigator Judgement | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Voluntary withdrawal | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event (AE) or Serious Adverse Event (SAE) | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 3 | 0 | 0 | 0 | 0
Period: RT Post Treatment Follow-up: Weeks 54-65
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen | Randomized Post-Treatment Follow-up Period: Placebo | Randomized Post-Treatment Follow-up Period: Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen
Started | 0 | 0 | 7 (Only those participants who were entered in the 13-week post-treatment follow-up period after the randomized treatment period.) | 9 (Only those participants who were entered in the 13-week post-treatment follow-up period after the randomized treatment period.) | 0 | 0
Completed | 0 | 0 | 6 | 7 | 0 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 0
Not completed — AE or SAE | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 2 | 0 | 0
Period: OLE Period-Year 1: Week 53 to 104
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen | Randomized Post-Treatment Follow-up Period: Placebo | Randomized Post-Treatment Follow-up Period: Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen
Started | 0 | 0 | 0 | 0 | 12 (Only those participants who were entered the in the OLE period (first OLE period) after the randomized treatment period.) | 12 (Only those participants who were entered the in the OLE period (first OLE period) after the randomized treatment period.)
Completed | 0 | 0 | 0 | 0 | 1 | 3
Not Completed | 0 | 0 | 0 | 0 | 11 | 9
Not completed — Investigator Judgement | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 3 | 1
Not completed — AE or SAE | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 5 | 7
Period: OLE Period-Year 2: Week 105 to 156
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen | Randomized Post-Treatment Follow-up Period: Placebo | Randomized Post-Treatment Follow-up Period: Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen
Started | 0 | 0 | 0 | 0 | 1 (Only those participants who were continuing the dosing for up to an additional 52 weeks in the second OLE period.) | 2 (Only those participants who were continuing the dosing for up to an additional 52 weeks in the second OLE period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 2
Period: PT Follow-up: Weeks 104 to 169
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen | Randomized Post-Treatment Follow-up Period: Placebo | Randomized Post-Treatment Follow-up Period: Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen
Started | 0 | 0 | 0 | 0 | 12 (Participants who were entered in the post-treatment follow-up after the OLE Period.) | 12 (Participants who were entered in the post-treatment follow-up after the OLE Period.)
Completed | 0 | 0 | 0 | 0 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Voluntary withdrawal | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least one dose of study drug in the randomized treatment period, and who had a baseline fasting triglyceride (TG) assessment.
Groups:
- Randomized Treatment Period: Placebo: Participants received volanesorsen-matching placebo as a SC injection once-weekly from Weeks 1 to 52 of the randomized treatment period. Participants were allowed dose adjustment based on monitoring rules
- Total: Total of all reporting groups
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12) | 46 (10) | 47 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 17 | 20 | 37
  Race: Asian | 1 | 1 | 2
  Race: Other Race | 1 | 0 | 1
Fasting Triglycerides [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 1290.95 (1296.19) | 1241.31 (1090.83) | 1264.89 (1177.40)
Hepatic Fat Fraction [Mean (Standard Deviation); unit: percentage (Hepatic Fat Fraction)] — Population: Number analyzed signifies the number of participants with data available for hepatic fat fraction.
  percentage (Hepatic Fat Fraction)
    number analyzed (Participants) | 16 | 17 | 33
    (all) | 17.00 (7.52) | 18.10 (8.41) | 17.57 (7.88)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.25 (1.13) | 7.84 (1.62) | 8.04 (1.40)
Short Form-36 (SF-36) Weighted Sum of Scores [Mean (Standard Deviation); unit: score on a scale] — The SF-36 Health Survey is a 36-item, patient-reported survey of patient health. SF-36 consists of 8 health dimensions,which are weighted sums of the questions in each section. SF-36 included 36 questions related to 8 health dimensions:physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning,emotional role functioning, and mental health. Each dimension was scored on a scale of 0 to 100 where, higher score = better quality of life. Population: Number analyzed signifies the number of participants with data available for SF-36 weighted sum of scores.
  score on a scale
    number analyzed (Participants) | 16 | 17 | 33
    (all) | 48.51 (12.83) | 46.31 (12.83) | 47.38 (12.45)
EQ-5D Questionnaires: Index Scores [Mean (Standard Deviation); unit: score on a scale] — EQ-5D-5L is a standardized health-related quality of life questionnaire. EQ-5D-5L consists of two components: a health state profile and VAS. EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state. Population: Number analyzed signifies the number of participants with data available for EQ-5D Questionnaires: Index Scores.
  score on a scale
    number analyzed (Participants) | 12 | 17 | 29
    (all) | 0.83 (0.20) | 0.84 (0.18) | 0.83 (0.19)
EQ-5D Questionnaires: Visual Analog Scale [Mean (Standard Deviation); unit: score on a scale] — EQ-5D-5L is a standardized health-related quality of life questionnaire EQ-5D-5L consists of two components: a health state profile and Visual Analog Scale (VAS). EQ-5D-5L- VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. Population: Number analyzed signifies the number of participants with data available for EQ-5D Questionnaires: VAS.
  score on a scale
    number analyzed (Participants) | 12 | 17 | 29
    (all) | 70 (18) | 71 (18) | 71 (17)

OUTCOME MEASURES:

1. Primary Outcome: Randomized Treatment Period: Percent Change From Baseline to Month 3 in Fasting Triglycerides (TG)
Description: Baseline was defined as the average of Day 1 predose fasting assessment and the last fasting measurement prior to Day 1 predose fasting assessment. Month 3 value was defined as the average of Week 12 and Week 13 fasting TG assessments of the randomized treatment period. The data was analyzed using an analysis of covariance (ANCOVA) model with the randomization stratification factor (diagnosis of disease with or without genetics and family history) and treatment group as factors and log-transformed baseline fasting TG as a covariate.
Time Frame: Baseline to Month 3
Population: FAS included all participants who were randomized and received at least one dose of study drug in the randomized treatment period, and who had a baseline fasting TG assessment. This outcome measure is reported here for the randomized treatment period only, as per the planned analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 21
percent change | -21.64 [-60.85 to 17.57] | -88.47 [-133.56 to -43.38]
Statistical Analysis 1: Comparison: Randomized Treatment Period: Placebo vs Randomized Treatment Period: Volanesorsen; Test type: Superiority; p = 0.0009, ANCOVA; Difference in Least Square Mean = -66.83, 95% CI 2-sided [-104.17 to -29.48]

2. Secondary Outcome: Randomized Treatment Period: Percent Change From Baseline in Hepatic Steatosis as Assessed by Hepatic Fat Fraction Using Magnetic Resonance Imaging (MRI)
Description: Baseline was defined as the last non-missing assessment prior to the first dose of study drug in the randomized treatment period. Randomized treatment period: Month 6 value was defined as Week 25 or Week 26 for MRI assessment and Month 12 was defined as Week 50 or Week 52 for MRI assessment. Hepatic steatosis is a reversible condition in which large vacuoles of triglyceride fat accumulate in the liver cells, causing nonspecific inflammation. Hepatic Steatosis was assessed by hepatic fat fraction using MRI.
Time Frame: Baseline, Months 6 and 12
Population: FAS included all participants who were randomized and received at least one dose of study drug in the randomized treatment period, and who had a baseline fasting TG assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 21
percent change
  Percent Change at Month 6 | 2.83 [-23.46 to 29.12] | -22.86 [-52.07 to 6.34]
  Percent Change at Month 12 | 1.46 [-30.49 to 33.42] | -51.87 [-87.87 to -15.87]
Statistical Analysis 1: Comparison: Randomized Treatment Period: Placebo vs Randomized Treatment Period: Volanesorsen; Month 6; Test type: Superiority; p = 0.0736, ANCOVA; Difference in Least Square Mean = -25.69, 95% CI 2-sided [-54.03 to 2.65]
Statistical Analysis 2: Comparison: Randomized Treatment Period: Placebo vs Randomized Treatment Period: Volanesorsen; Month 12; Test type: Superiority; p = 0.0039, ANCOVA; Difference in Least Square Mean = -53.33, 95% CI 2-sided [-87.71 to -18.95]

3. Secondary Outcome: Open-Label Extension Period: Percent Change From Baseline in Hepatic Steatosis as Assessed by Hepatic Fat Fraction Using MRI
Description: Baseline was defined as the last non-missing assessment prior to the first dose of study drug in the randomized treatment period. Open-label extension period: Month 6 value was defined as Week 77 or Week 78 for MRI assessment and Month 12 value was defined as Week 102 or Week 104 for MRI assessment. Hepatic steatosis is a reversible condition in which large vacuoles of triglyceride fat accumulate in the liver cells, causing nonspecific inflammation. Hepatic Steatosis was assessed by hepatic fat fraction using MRI.
Time Frame: Baseline, Months 6 and 12
Population: FAS included all participants who were randomized and received at least one dose of study drug in the open-label extension period, and who had a baseline fasting TG assessment. Here, "number analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Open-Label Extension Period: Placebo/Volanesorsen: Participants in the Randomized Treatment Period: Placebo arm group who completed the randomized treatment period, were to receive 300 mg of volanesorsen as a SC injection once-weekly for 52 weeks (from Weeks 53 to 104) in the OLE period. Participants were allowed dose adjustment based on monitoring rules. After Week 104 of the OLE period, participants had the option of continuing treatment with 300 mg of volanesorsen as a SC injection for up to an additional 52 weeks (from Week 105 to 156).
- Open-Label Extension Period: Volanesorsen/Volanesorsen: Participants in the Randomized Treatment Period: Volanesorsen arm group who completed the randomized treatment period, received 300 mg of volanesorsen as a SC injection once-weekly for 52 weeks (from Weeks 53 to 104) in the OLE period. Participants were allowed dose adjustment based on monitoring rules. After Week 104 of the OLE period, participants had the option of continuing treatment with 300 mg of volanesorsen as a SC injection for up to an additional 52 weeks (from Week 105 to 156).
Arm/Group | Open-Label Extension Period: Placebo/Volanesorsen | Open-Label Extension Period: Volanesorsen/Volanesorsen
Number analyzed (Participants) | 12 | 12
percent change
  Percent Change at Month 6: number analyzed (Participants) | 6 | 5
  Percent Change at Month 6 | -18.4 (54.7) | -60.2 (43.6)
  Percent Change at Month 12: number analyzed (Participants) | 2 | 2
  Percent Change at Month 12 | -93.5 (44.4) | -22.1 (47.5)

4. Secondary Outcome: Randomized Treatment Period: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: Baseline was defined as the last non-missing assessment prior to the first dose of study drug. Randomized treatment period: The Month 3 value was defined as Week 13, Month 6 value was defined as Week 26, Month 9 value was defined as Week 38 and Month 12 value was defined as Week 52.
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 21
percentage of HbA1c
  Change at Month 3 | -0.51 [-1.22 to 0.20] | -0.21 [-1.00 to 0.58]
  Change at Month 6 | 0.06 [-1.02 to 1.15] | 0.26 [-0.98 to 1.50]
  Change at Month 9 | 0.68 [-0.49 to 1.85] | 0.48 [-0.84 to 1.80]
  Change at Month 12 | 0.48 [-0.49 to 1.45] | 0.28 [-0.78 to 1.35]
Statistical Analysis 1: Comparison: Randomized Treatment Period: Placebo vs Randomized Treatment Period: Volanesorsen; Month 3; Test type: Superiority; p = 0.4108, ANCOVA; Difference in Least Square Mean = 0.30, 95% CI 2-sided [-0.43 to 1.03]
Statistical Analysis 2: Comparison: Randomized Treatment Period: Placebo vs Randomized Treatment Period: Volanesorsen; Month 6; Test type: Superiority; p = 0.7308, ANCOVA; Difference in Least Square Mean = 0.19, 95% CI 2-sided [-0.95 to 1.34]
Statistical Analysis 3: Comparison: Randomized Treatment Period: Placebo vs Randomized Treatment Period: Volanesorsen; Month 9; Test type: Superiority; p = 0.7511, ANCOVA; Difference in Least Square Mean = -0.20, 95% CI 2-sided [-1.45 to 1.06]
Statistical Analysis 4: Comparison: Randomized Treatment Period: Placebo vs Randomized Treatment Period: Volanesorsen; Month 12; Test type: Superiority; p = 0.7659, ANCOVA; Difference in Least Square Mean = -0.19, 95% CI 2-sided [-1.52 to 1.13]

5. Secondary Outcome: Open Label Extension Period: Change From Baseline in HbA1c
Description: Baseline was defined as the last non-missing assessment prior to the first dose of study drug. Open-label extension period: Month 3 value was defined as Week 65, Month 6 value was defined as Week 78, Month 9 value was defined as Week 90 and Month 12 value was defined as Week 104.
Time Frame: Baseline, Months 3, 6, 9, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Open-Label Extension Period: Placebo/Volanesorsen | Open-Label Extension Period: Volanesorsen/Volanesorsen
Number analyzed (Participants) | 12 | 12
percentage of HbA1c
  Change at Month 3: number analyzed (Participants) | 6 | 8
  Change at Month 3 | 0.42 (1.54) | 0.91 (2.18)
  Change at Month 6: number analyzed (Participants) | 6 | 3
  Change at Month 6 | 0.35 (1.54) | -0.75 (0.35)
  Change at Month 9: number analyzed (Participants) | 2 | 2
  Change at Month 9 | 0.35 (1.06) | -0.05 (0.64)
  Change at Month 12: number analyzed (Participants) | 2 | 2
  Change at Month 12 | 0.00 (0.71) | 0.30 (0.99)

6. Secondary Outcome: Randomized Treatment Period: Percentage of Participants Who Achieved Greater Than or Equal to (≥) 40% Reduction in Fasting Triglyceride and ≥ 30% Reduction of Hepatic Fat Fraction at Month 6
Description: The baseline of TG is defined as the average of Day 1 pre-dose fasting assessment and the last fasting measurement prior to Day 1 pre-dose fasting assessment. The baseline of hepatic fat fraction is defined as the last non-missing assessment prior to the first dose of study drug. Randomized treatment period: Month 6 value was defined as average of Week 25 and Week 26 for fasting TG and Week 25 or Week 26 for hepatic fat fraction.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 21
percentage of participants | 5.3 | 42.9

7. Secondary Outcome: Randomized Treatment Period: Change From Baseline in Disease Burden Score
Description: The Disease Burden Score is a questionnaire that allows participants to self-report their chronic conditions and then assess the degree to which each condition interferes with daily activities.
Time Frame: From the first dose of study drug to Week 52
Population: Data for this outcome measure was not collected due to the change in planned analysis.
Groups:
- Randomized Treatment Period: Placebo: Participants received volanesorsen-matching placebo as a SC injection once weekly from Weeks 1 to 52 of the randomized treatment period. Participants were allowed dose adjustment based on monitoring rules.
- Randomized Treatment Period: Volanesorsen: Participants received 300 mg of volanesorsen as a SC injection once weekly from Weeks 1 to 52 of the randomized treatment period. Participants were allowed dose adjustment based on monitoring rules.
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Open-Label Extension Period: Change From Baseline in Disease Burden Score
Description: as for outcome 7
Time Frame: From the first dose of study drug in open label extension period to Week 117
Population: Data for this outcome measure was not collected due to the change in planned analysis.
Arm/Group | Open-Label Extension Period: Placebo/Volanesorsen | Open-Label Extension Period: Volanesorsen/Volanesorsen
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Randomized Treatment Period: Patient-Reported Pain
Description: Patient-reported pain was assessed by rating pain symptoms at its worst and least for the last 24 hours, on average, and at the moment, with 0 as the lowest score (no pain) and 10 as the highest score (worst pain as you can imagine). Patient-reported pain was also assessed by rating pain symptoms (rate pain on average, rate pain right now) that interfered with general activity, interfered with mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life, with 0 as the lowest score (did not interfered) and 10 as the highest score (completely interfered). The scores from each assessment time point were averaged for all of the below reported categories.
Time Frame: From the first dose of study drug up to Week 52
Population: FAS included all participants who were randomized and received at least one dose of study drug in the randomized treatment period, and who had a baseline fasting TG assessment. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 20
score on a scale
  Rate Pain at its Worst Last 24 Hours | 3.28 (2.79) | 3.57 (2.72)
  Rate Pain at its Least Last 24 Hours | 2.45 (2.46) | 2.59 (2.43)
  Rate Pain on Average | 3.08 (2.62) | 3.16 (2.47)
  Rate Pain Right Now | 2.72 (2.59) | 2.96 (2.50)
  General Activity | 2.43 (2.80) | 2.83 (2.57)
  Interfere With Mood | 2.31 (2.88) | 2.98 (2.59)
  Walking Ability | 2.35 (2.96) | 2.79 (2.59)
  Normal Work | 2.37 (2.84) | 2.89 (2.56)
  Relations With Other People | 2.23 (2.79) | 2.62 (2.67)
  Sleep | 2.75 (2.95) | 2.73 (2.75)
  Enjoyment of Life | 2.42 (2.82) | 2.68 (2.62)

10. Secondary Outcome: Open Label Extension Period: Patient-Reported Pain
Description: as for outcome 9
Time Frame: From the first dose of study drug in open label extension period up to Week 117
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Extension Period: Placebo/Volanesorsen | Open-Label Extension Period: Volanesorsen/Volanesorsen
Number analyzed (Participants) | 9 | 9
score on a scale
  Rate Pain at its Worst Last 24 Hours | 1.70 (1.18) | 3.82 (2.97)
  Rate Pain at its Least Last 24 Hours | 0.95 (1.04) | 2.78 (2.60)
  Rate Pain on Average | 1.35 (1.22) | 3.16 (2.72)
  Rate Pain Right Now | 1.28 (1.18) | 3.49 (2.99)
  General Activity | 1.03 (1.45) | 3.28 (2.90)
  Interfere With Mood | 1.27 (1.46) | 3.23 (2.94)
  Walking Ability | 1.05 (1.50) | 3.51 (2.83)
  Normal Work | 1.08 (1.40) | 3.48 (2.98)
  Relations With Other People | 1.08 (1.48) | 3.18 (3.09)
  Sleep | 1.51 (1.83) | 3.13 (3.35)
  Enjoyment of Life | 1.23 (1.65) | 3.33 (2.94)

11. Secondary Outcome: Randomized Treatment Period: Patient-Reported Hunger
Description: Patient-reported hunger was assessed by participants who completed a questionnaire about: how hungry you feel, how satisfied you feel, how full you feel, how much you think you can eat, like to eat something sweet, like to eat something salty, like to eat something savory and like to eat something fatty. Participants also rated the palatability of meals that included visual appeal, smell, taste, and aftertaste. Scores of 1-39 were categorized as mild, 40-69 as moderate, and 70-100 as severe. The scores from each assessment time point were averaged for all of the below reported categories.
Time Frame: From the first dose of study drug up to Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 20
score on a scale
  How Hungry You Feel | 29.4 (20.7) | 29.6 (14.4)
  How Satisfied You Feel | 56.8 (22.4) | 57.5 (15.1)
  How Full You Feel | 62.6 (20.5) | 56.6 (18.4)
  How Much You Think You Can Eat | 33.6 (22.1) | 36.8 (15.4)
  Like to Eat Something Sweet | 71.0 (20.8) | 54.8 (27.1)
  Like to Eat Something Salty | 66.9 (21.7) | 69.0 (20.2)
  Like to Eat Something Savory | 65.2 (21.4) | 66.8 (21.9)
  Like to Eat Something Fatty | 77.9 (18.4) | 75.9 (22.2)
  Visual Appeal | 28.6 (20.5) | 34.5 (21.0)
  Smell | 23.4 (16.2) | 25.4 (15.5)
  Taste | 25.5 (18.3) | 29.1 (14.5)
  Aftertaste | 58.9 (27.5) | 51.0 (24.6)
  Palatability | 31.3 (20.1) | 32.2 (15.1)

12. Secondary Outcome: Open Label Extension Period: Patient-Reported Hunger
Description: as for outcome 11
Time Frame: From the first dose of study drug in open label extension period up to Week 117
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Open-Label Extension: Volanesorsen/Volanesorsen: Participants in the Randomized Treatment Period: Volanesorsen arm group who completed the randomized treatment period, received 300 mg of volanesorsen as a SC injection once-weekly for 52 weeks (from Weeks 53 to 104) in the OLE period. Participants were allowed dose adjustment based on monitoring rules. After Week 104 of the OLE period, participants had the option of continuing treatment with 300 mg of volanesorsen as a SC injection for up to an additional 52 weeks (from Week 105 to 156).
Arm/Group | Open-Label Extension Period: Placebo/Volanesorsen | Open-Label Extension: Volanesorsen/Volanesorsen
Number analyzed (Participants) | 9 | 9
score on a scale
  How Hungry You Feel | 29.9 (23.3) | 33.2 (23.2)
  How Satisfied You Feel | 54.2 (23.3) | 56.3 (20.2)
  How Full You Feel | 59.7 (22.2) | 52.9 (24.4)
  How Much You Think You Can Eat | 34.0 (21.8) | 34.9 (21.5)
  Like to Eat Something Sweet | 73.7 (25.4) | 57.9 (24.0)
  Like to Eat Something Salty | 65.7 (28.1) | 61.9 (22.1)
  Like to Eat Something Savory | 65.4 (24.7) | 62.7 (30.5)
  Like to Eat Something Fatty | 80.7 (18.1) | 68.0 (30.4)
  Visual Appeal | 14.9 (16.1) | 35.3 (25.9)
  Smell | 13.1 (14.3) | 29.6 (21.6)
  Taste | 13.6 (15.1) | 32.9 (25.0)
  Aftertaste | 48.1 (38.6) | 56.9 (29.3)
  Palatability | 24.4 (23.4) | 37.3 (20.6)

13. Secondary Outcome: Randomized Treatment Period: Change From Baseline in Mean Short Form-36 (SF-36) Weighted Sum of Scores
Description: The SF-36 Health Survey is a 36-item, patient-reported survey of patient health. SF-36 consists of 8 health dimensions,which are weighted sums of the questions in each section. SF-36 included 36 questions related to 8 health dimensions:physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning,emotional role functioning, and mental health. Each dimension was scored on a scale of 0 to 100 where, higher score = better quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 13, 26 and 52
Population: FAS included all participants who were randomized and received at least one dose of study drug in the randomized treatment period, and who had a baseline fasting TG assessment. Here, "number analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 21
score on a scale
  Vitality: Change at Week 13: number analyzed (Participants) | 13 | 14
  Vitality: Change at Week 13 | -1.14 (7.33) | -0.21 (5.64)
  Vitality: Change at Week 26: number analyzed (Participants) | 12 | 15
  Vitality: Change at Week 26 | -0.25 (9.00) | -0.79 (6.89)
  Vitality: Change at Week 52: number analyzed (Participants) | 7 | 9
  Vitality: Change at Week 52 | -0.85 (6.11) | -3.30 (8.20)
  Physical Functioning: Change at Week 13: number analyzed (Participants) | 13 | 14
  Physical Functioning: Change at Week 13 | -0.29 (4.81) | -0.41 (3.91)
  Physical Functioning: Change at Week 26: number analyzed (Participants) | 12 | 15
  Physical Functioning: Change at Week 26 | -0.64 (6.49) | 0.51 (5.29)
  Physical Functioning: Change at Week 52: number analyzed (Participants) | 7 | 9
  Physical Functioning: Change at Week 52 | -3.55 (4.05) | -2.76 (5.25)
  Bodily Pain: Change at Week 13: number analyzed (Participants) | 13 | 14
  Bodily Pain: Change at Week 13 | -0.46 (7.97) | 0.75 (6.26)
  Bodily Pain: Change at Week 26: number analyzed (Participants) | 12 | 15
  Bodily Pain: Change at Week 26 | -1.98 (12.24) | 0.19 (4.27)
  Bodily Pain: Change at Week 52: number analyzed (Participants) | 7 | 9
  Bodily Pain: Change at Week 52 | -0.29 (6.35) | -2.55 (8.48)
  General Health Perceptions: Change at Week 13: number analyzed (Participants) | 13 | 14
  General Health Perceptions: Change at Week 13 | -0.55 (5.57) | -0.58 (4.04)
  General Health Perceptions: Change at Week 26: number analyzed (Participants) | 12 | 15
  General Health Perceptions: Change at Week 26 | -1.59 (5.00) | 0.54 (7.25)
  General Health Perceptions: Change at Week 52: number analyzed (Participants) | 7 | 9
  General Health Perceptions: Change at Week 52 | -1.50 (6.74) | -1.48 (4.53)
  Physical Role Functioning: Change at Week 13: number analyzed (Participants) | 13 | 14
  Physical Role Functioning: Change at Week 13 | -0.52 (5.44) | -0.64 (4.61)
  Physical Role Functioning: Change at Week 26: number analyzed (Participants) | 12 | 15
  Physical Role Functioning: Change at Week 26 | -2.06 (10.81) | 0.75 (4.70)
  Physical Role Functioning: Change at Week 52: number analyzed (Participants) | 7 | 9
  Physical Role Functioning: Change at Week 52 | -0.32 (2.02) | -2.00 (7.05)
  Emotional Role Functioning: Change at Week 13: number analyzed (Participants) | 13 | 14
  Emotional Role Functioning: Change at Week 13 | -1.88 (4.63) | 0.75 (6.85)
  Emotional Role Functioning: Change at Week 26: number analyzed (Participants) | 12 | 15
  Emotional Role Functioning: Change at Week 26 | -2.90 (6.44) | 0.23 (7.50)
  Emotional Role Functioning : Change at Week 52: number analyzed (Participants) | 7 | 9
  Emotional Role Functioning : Change at Week 52 | -1.00 (5.94) | -5.42 (5.80)
  Social Role Functioning: Change at Week 13: number analyzed (Participants) | 13 | 14
  Social Role Functioning: Change at Week 13 | -3.86 (9.85) | 1.07 (4.02)
  Social Role Functioning: Change at Week 26: number analyzed (Participants) | 12 | 15
  Social Role Functioning: Change at Week 26 | -5.01 (9.07) | -0.67 (3.21)
  Social Role Functioning: Change at Week 52: number analyzed (Participants) | 7 | 9
  Social Role Functioning: Change at Week 52 | 2.87 (4.89) | -2.79 (7.14)
  Mental Health: Change at Week 13: number analyzed (Participants) | 13 | 14
  Mental Health: Change at Week 13 | 0.00 (6.67) | -0.19 (7.91)
  Mental Health: Change at Week 26: number analyzed (Participants) | 12 | 15
  Mental Health: Change at Week 26 | -2.18 (7.71) | 1.05 (6.76)
  Mental Health: Change at Week 52: number analyzed (Participants) | 7 | 9
  Mental Health: Change at Week 52 | -0.37 (6.66) | -1.75 (6.13)

14. Secondary Outcome: Open-Label Extension Period: Change From Baseline in Mean SF-36 Weighted Sum of Scores
Description: as for outcome 13
Time Frame: Baseline, Weeks 65, 78 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Extension Period: Placebo/Volanesorsen | Open-Label Extension Period: Volanesorsen/Volanesorsen
Number analyzed (Participants) | 12 | 12
score on a scale
  Vitality: Change at Week 65: number analyzed (Participants) | 2 | 7
  Vitality: Change at Week 65 | 4.46 (6.30) | -0.42 (13.88)
  Vitality: Change at Week 78: number analyzed (Participants) | 2 | 1
  Vitality: Change at Week 78 | -2.98 (12.61) | -2.97 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Vitality: Change at Week 104: number analyzed (Participants) | 1 | 1
  Vitality: Change at Week 104 | 2.97 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -5.94 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Physical Functioning: Change at Week 65: number analyzed (Participants) | 2 | 7
  Physical Functioning: Change at Week 65 | -4.79 (6.77) | -1.37 (5.81)
  Physical Functioning: Change at Week 78: number analyzed (Participants) | 2 | 1
  Physical Functioning: Change at Week 78 | -3.83 (5.41) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Physical Functioning: Change at Week 104: number analyzed (Participants) | 1 | 1
  Physical Functioning: Change at Week 104 | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.91 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Bodily Pain: Change at Week 65: number analyzed (Participants) | 2 | 7
  Bodily Pain: Change at Week 65 | -2.42 (3.42) | 0.40 (7.13)
  Bodily Pain: Change at Week 78: number analyzed (Participants) | 2 | 1
  Bodily Pain: Change at Week 78 | -7.26 (19.39) | -11.29 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Bodily Pain: Change at Week 104: number analyzed (Participants) | 1 | 1
  Bodily Pain: Change at Week 104 | 6.45 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -10.49 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  General Health Perceptions: Change at Week 65: number analyzed (Participants) | 2 | 7
  General Health Perceptions: Change at Week 65 | 2.38 (3.36) | -2.38 (4.42)
  General Health Perceptions: Change at Week 78: number analyzed (Participants) | 2 | 1
  General Health Perceptions: Change at Week 78 | -2.86 (7.40) | -4.75 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  General Health Perceptions: Change at Week 104: number analyzed (Participants) | 1 | 1
  General Health Perceptions: Change at Week 104 | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -4.75 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Physical Role Functioning: Change at Week 65: number analyzed (Participants) | 2 | 7
  Physical Role Functioning: Change at Week 65 | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0 (6.22)
  Physical Role Functioning: Change at Week 78: number analyzed (Participants) | 2 | 1
  Physical Role Functioning: Change at Week 78 | -10.11 (14.29) | -2.25 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Physical Role Functioning: Change at Week 104: number analyzed (Participants) | 1 | 1
  Physical Role Functioning: Change at Week 104 | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -4.50 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Emotional Role Functioning: Change at Week 65: number analyzed (Participants) | 2 | 7
  Emotional Role Functioning: Change at Week 65 | -1.74 (2.46) | -3.48 (11.37)
  Emotional Role Functioning: Change at Week 78: number analyzed (Participants) | 2 | 1
  Emotional Role Functioning: Change at Week 78 | 1.74 (2.46) | -10.45 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Emotional Role Functioning: Change at Week 104: number analyzed (Participants) | 1 | 1
  Emotional Role Functioning: Change at Week 104 | 3.48 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -10.45 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Social Role Functioning: Change at Week 65: number analyzed (Participants) | 2 | 7
  Social Role Functioning: Change at Week 65 | 5.02 (7.09) | -2.15 (7.58)
  Social Role Functioning: Change at Week 78: number analyzed (Participants) | 2 | 1
  Social Role Functioning: Change at Week 78 | -2.15 (7.09) | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Social Role Functioning: Change at Week 104: number analyzed (Participants) | 1 | 1
  Social Role Functioning: Change at Week 104 | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Mental Health: Change at Week 65: number analyzed (Participants) | 2 | 7
  Mental Health: Change at Week 65 | -5.23 (11.10) | -1.12 (13.67)
  Mental Health: Change at Week 78: number analyzed (Participants) | 2 | 1
  Mental Health: Change at Week 78 | 6.54 (9.25) | -15.70 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Mental Health: Change at Week 104: number analyzed (Participants) | 1 | 1
  Mental Health: Change at Week 104 | 2.62 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable.

15. Secondary Outcome: Randomized Treatment Period: Change From Baseline in Mean EQ-5D: Index Scores and Visual Analog Scale (VAS)
Description: EQ-5D-5L is a standardized health-related quality of life questionnaire developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L consists of two components: a health state profile and VAS. EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state. EQ-5D-5L- VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A negative change from baseline indicates worsening. A positive change from baseline indicates improvement.
Time Frame: Baseline, Weeks 13, 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen
Number analyzed (Participants) | 19 | 21
score on a scale
  Index Score: Change at Week 13: number analyzed (Participants) | 8 | 14
  Index Score: Change at Week 13 | 0.05 (0.10) | -0.02 (0.06)
  Index Score: Change at Week 26: number analyzed (Participants) | 9 | 15
  Index Score: Change at Week 26 | -0.11 (0.19) | -0.02 (0.12)
  Index Score: Change at Week 52: number analyzed (Participants) | 4 | 9
  Index Score: Change at Week 52 | -0.08 (0.10) | -0.05 (0.07)
  EQ VAS Score: Change at Week 13: number analyzed (Participants) | 8 | 14
  EQ VAS Score: Change at Week 13 | -2 (13) | -2 (15)
  EQ VAS Score: Change at Week 26: number analyzed (Participants) | 9 | 15
  EQ VAS Score: Change at Week 26 | -11 (17) | -2 (14)
  EQ VAS Score: Change at Week 52: number analyzed (Participants) | 4 | 9
  EQ VAS Score: Change at Week 52 | -13 (18) | -4 (16)

16. Secondary Outcome: Open-Label Extension Period: Change From Baseline in Mean EQ-5D: Index and Visual Analog Scale (VAS) Scores
Description: as for outcome 15
Time Frame: Baseline, Weeks 65, 78 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Extension Period: Placebo/Volanesorsen | Open-Label Extension Period: Volanesorsen/Volanesorsen
Number analyzed (Participants) | 12 | 12
score on a scale
  Index Score: Change at Week 65: number analyzed (Participants) | 0 | 7
  Index Score: Change at Week 65 |  | -0.06 (0.08)
  Index Score: Change at Week 78: number analyzed (Participants) | 2 | 1
  Index Score: Change at Week 78 | -0.02 (0.03) | -0.07 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Index Score: Change at Week 104: number analyzed (Participants) | 1 | 1
  Index Score: Change at Week 104 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.27 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EQ VAS Score: Change at Week 65: number analyzed (Participants) | 0 | 7
  EQ VAS Score: Change at Week 65 |  | -4 (16)
  EQ VAS Score: Change at Week 78: number analyzed (Participants) | 2 | 1
  EQ VAS Score: Change at Week 78 | -15 (22) | -6 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EQ VAS Score: Change at Week 104: number analyzed (Participants) | 1 | 1
  EQ VAS Score: Change at Week 104 | 2 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable.

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of follow-up period [Up to Week 169]
Description: Safety Population Set 1 included all participants who were randomized and received at least one dose of study drug (volanesorsen or placebo) in the randomized treatment period. Safety Population Set 2 included all participants who entered the OLE Period and received at least one dose of study drug (volanesorsen) in the OLE period.
Groups:
- Randomized Post-Treatment Follow-up: Placebo: Following the randomized treatment period, participants who received volanesorsen-matching placebo in randomized treatment period and did not enter the OLE period went straight to the 13-week post-treatment follow-up period.
- Randomized Post-Treatment Follow-up: Volanesorsen: Following the randomized treatment period, participants who received 300 mg of volanesorsen in randomized treatment period and did not enter in the OLE period went straight to the 13-week post-treatment follow-up period.
Arm/Group | Randomized Treatment Period: Placebo | Randomized Treatment Period: Volanesorsen | Randomized Post-Treatment Follow-up: Placebo | Randomized Post-Treatment Follow-up: Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/7 | 0/9 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/19 | 6/21 | 1/7 | 1/9 | 4/12 | 4/12
Other Adverse Events (participants affected / at risk) | 18/19 | 21/21 | 4/7 | 5/9 | 11/12 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Treatment Period: Placebo (N=19) | Randomized Treatment Period: Volanesorsen (N=21) | Randomized Post-Treatment Follow-up: Placebo (N=7) | Randomized Post-Treatment Follow-up: Volanesorsen (N=9) | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen (N=12) | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Medical device site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Treatment Period: Placebo (N=19) | Randomized Treatment Period: Volanesorsen (N=21) | Randomized Post-Treatment Follow-up: Placebo (N=7) | Randomized Post-Treatment Follow-up: Volanesorsen (N=9) | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Placebo/Volanesorsen (N=12) | Open-Label Extension Period (OLE and OLE Post-Treatment Follow-up): Volanesorsen/Volanesorsen (N=12)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 1 | 0 | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 0 | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 6 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 13 | 0 | 0 | 7 | 1
Injection site pruritus (General disorders) | 0 | 11 | 0 | 0 | 3 | 0
Injection site pain (General disorders) | 3 | 7 | 0 | 0 | 4 | 1
Injection site swelling (General disorders) | 0 | 8 | 0 | 0 | 6 | 2
Fatigue (General disorders) | 3 | 2 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 3 | 0 | 0 | 3 | 0
Injection site reaction (General disorders) | 0 | 3 | 0 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 3 | 0 | 0 | 2 | 0
Injection site mass (General disorders) | 0 | 3 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 2 | 0 | 0 | 1 | 0
Injection site nodule (General disorders) | 0 | 2 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 2 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 3 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Injection site warmth (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 3 | 0 | 0 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epulis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 5 | 0 | 0 | 2 | 2
Haemoglobin decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 1
Protein total increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 2
Cardiac murmur (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Blood glucose fluctuation (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Glucose urine (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Red blood cells urine (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Urine protein, quantitative (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Synovial fluid white blood cells positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Rheumatoid factor increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Echocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Biopsy muscle (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Bacterial test (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Albumin urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 4 | 0 | 0 | 3 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysstasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Splinter (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sleep-related eating disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnambulism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Muscular dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthma prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Microcytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The Sponsor decided to terminate the study early at a time point when sufficient data had been accumulated to inform a decision on further development of volanesorsen in participants with FPL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT02527343/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT02527343/SAP_001.pdf